CLINICAL TRIAL: NCT06958354
Title: Evaluation of the Clinical Relationship Between Procalcitonin Level and Bacteremia Agent in Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mete Erdemir, specialist, Gulhane Training and Research Hospital
Other Study IDs: 2023/34
Record Dates: First submitted 2025-04-24; First posted 2025-05-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-04

CONDITIONS: Sepsis; Septic; Bacteremia and Sepsis; Intensive Care Medicine; Procalcitonin
Keywords: procalcitonin; sepsis; septic shock; intrensive care medicine
MeSH Terms: conditions — Sepsis; Bacteremia; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

SUMMARY:
In intensive care units, sepsis, which can be defined as bacteremia and the irregular and uncontrolled inflammatory response to it, is one of the most important causes of mortality. Early recognition of sepsis and appropriate antibiotic use for the causative agent is one of the most important steps in the fight against sepsis. Procalcitonin (PCT) is a calcitonin precursor peptide and has been reported to predict bacteremia early. While the PCT concentration level is negligible in healthy individuals, it has been shown to increase especially in bacterial infections, sepsis, trauma and burns. In our study, our aim is to determine whether there is a relationship between serum PCT concentration levels taken within 24 hours according to the time of the sample taken for blood culture with growth in patients followed up in our Internal Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Positive blood culture during their follow up
* Patients over 18 years of age

Exclusion Criteria:

* Those under the age of 18
* Those who have had surgery or trauma in the last 72 hours
* Those with a history of autoimmune disease, chronic renal failure
* Patients admitted to intensive care due to acute pancreatitis, pregnancy, burns.
* Patients with incomplete data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Among the patients who were followed up in the intensive care unit between 01.01.2018 and 01.01.2023 and who were found to have a positive blood culture during their follow up, only those whose PCT results were obtained within 24 hours, based on the time the blood culture sample was taken, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1529 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-10-19 (Actual)

PRIMARY OUTCOMES:
Correlation of serum PCT levels measured within 24 hours of culture in intensive care patients with bacteremia and the pathogen type (Gram-positive, Gram-negative, fungal) in the culture result. | In patients with positive blood cultures, serum PCT values studied within the first 24 hours from the time the culture sample was taken will be evaluated retrospectively.

SECONDARY OUTCOMES:
Diagnostic power of PCT levels in distinguishing Gram-negative, Gram-positive and fungal infections | serum PCT values studied within the first 24 hours from the time the culture sample

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data to be Shared:
  Anonymized individual patient data (demographic information, laboratory results, culture results, clinical scores and mortality status).
  Sharing Time:
  After the study is completed and the results are published
  Sharing Conditions:
  Requests with ethics committee approval and scientific purposes will be evaluated with a written application. Data sharing will be done via e-mail or secure systems by signing a data usage protocol.
  Sharing Scope:
  Only anonymous data will be shared, excluding identifying personal information
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Muller F, Christ-Crain M, Bregenzer T, Krause M, Zimmerli W, Mueller B, Schuetz P; ProHOSP Study Group. Procalcitonin levels predict bacteremia in patients with community-acquired pneumonia: a prospective cohort trial. Chest. 2010 Jul;138(1):121-9. doi: 10.1378/chest.09-2920. Epub 2010 Mar 18. PMID 20299634
- [Background] Liu D, Su L, Han G, Yan P, Xie L. Prognostic Value of Procalcitonin in Adult Patients with Sepsis: A Systematic Review and Meta-Analysis. PLoS One. 2015 Jun 15;10(6):e0129450. doi: 10.1371/journal.pone.0129450. eCollection 2015. PMID 26076027
- [Background] Leli C, Ferranti M, Moretti A, Al Dhahab ZS, Cenci E, Mencacci A. Procalcitonin levels in gram-positive, gram-negative, and fungal bloodstream infections. Dis Markers. 2015;2015:701480. doi: 10.1155/2015/701480. Epub 2015 Mar 17. PMID 25852221
- [Background] https://pmc.ncbi.nlm.nih.gov/articles/PMC6289022/